CLINICAL TRIAL: NCT04325815
Title: Multi-Centre, Open-label, Randomised, Prospective Trial to Assess Efficacy and Safety of the CADDIE Artificial Intelligence System for Improving Endoscopic Detection of Colonic Polyps in Real-time.
Brief Title: CADDIE Trial - Computer Aided Diagnosis and Detection for Intelligent Endoscopy
Acronym: CADDIE
Status: Completed | Type: Observational
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Other Study IDs: 126166
Record Dates: First submitted 2020-03-11; First posted 2020-03-30 (Actual); Results first posted 2025-02-19 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Polyps; Adenoma Colon; Colorectal Polyp; Colon Polyp
Keywords: Artificial Intelligence; Endoscopy; ADR
MeSH Terms: conditions — Polyps; Colonic Polyps | interventions — Endoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CADDIE: The endoscopist will be assisted with CADDIE system to detect polyps. The endoscopist will perform optical diagnosis of polyps with the assistance of the CADDIE's polyp characterisation function.
  Interventions: Device: CADDIE- Computer Aided (AI) Device used in Endoscopy
- Standard Procedure: In addition to routine colonoscopy the endoscopist will perform optical diagnosis of detected polyps without the assistance of the CADDIE.

INTERVENTIONS:
Device: CADDIE- Computer Aided (AI) Device used in Endoscopy — 1. CADDIE assisted polyp detection
  2. CADDIE assisted polyp characterisation
  Groups: CADDIE

SUMMARY:
Background:

Colonoscopy is accepted to be the gold standard for screening of colorectal cancer (CRC). Most CRCs develop from adenomatous polyps, with colonoscopy accepted to be the gold standard for screening of CRC. An endoscopist's ability to detect polyps is assessed in the form of an Adenoma Detection Rate (ADR). Each 1.0% increase in ADR is associated with a 3.0% decrease in the risk of the patient developing an interval CRC. There remains a wide variation in endoscopist ADR.

More recently, the use of artificial intelligence (AI) and computer aided diagnosis in endoscopy has been gaining increasing attention for its role in automated lesion detection and characterisation. AI can potentially improve ADR, but previous AI related work has largely focused on retrospectively assessing still endoscopic images and selected video sequences which may be subject to bias and lack clinical utility. There are only limited clinical studies evaluating the effect of AI in improving ADR.

The CADDIE device uses convolutional neural networks developed for computer assisted detection and computer assisted diagnosis of polyps.

Primary objective: To determine whether the CADDIE artificial intelligence system improves endoscopic detection of adenomas during colonoscopy.

Primary endpoint: The difference in adenoma detection rate (ADR) between the intervention (supported with the CADDIE system) and non-intervention arm

Study design: Multi-Centre, open-label, randomised, prospective trial to assess efficacy and safety of the CADDIE artificial intelligence system for improving endoscopic detection of colonic polyps in real-time.

ELIGIBILITY:
Inclusion Criteria:

* Patient's scheduled to undergo a surveillance or symptomatic colonoscopy with an endoscopist participating in the study phase of the trial.
* Male and female participants aged 18 years or older at the time of informed consent.
* Patient's able to comprehend, sign and date the written informed consent document to participate in the study.

Exclusion Criteria:

* Emergency colonoscopies and/or inpatient colonoscopies.
* Patients with inflammatory bowel disease (IBD)
* Patients with Colorectal Cancer (CRC)
* Patients with previous CRC
* Patients with previous colonic resection
* Patients returning for a planned elective therapeutic colonoscopy.
* Polyposis syndromes
* Current or relevant history of a physical or psychiatric illness or any medical condition that in the opinion of the investigator could affect the patient's safety or interfere with the study assessments
* Patients with a contraindication for biopsy or polypectomy. These include:

  * Patients who have not withheld medications pre-disposing to bleeding at time of colonoscopy as per local site /national guidelines 30.
  * Patients with a history of haemostasis disorders (Haemostasis disorders will include but will not be limited to: patients with haemophilia or other congenitally acquired clotting factor deficiencies, patients with cirrhosis with coagulopathy, patients known to have thrombocytopenia (<80,000 platelet/ul) and individuals with Von Willebrand's disease or other known platelet malfunction disorders).
* Patients is enrolled in another research study with an investigational medicinal product (IMP) or non-IMP that pre-disposes them to bleeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population will include patient's scheduled to undergo a surveillance or symptomatic colonoscopy at the participating sites.
Sampling Method: Non-Probability Sample
Enrollment: 739 (Actual)
Dates: Start 2021-04-29 (Actual); Primary Completion 2023-03-08 (Actual); Study Completion 2023-03-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manish Chand, MBBS FRCS PhD, Principal Investigator — UCL
Locations (1):
- University College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Patients will be asked informed consent with the possibility to share the data
Time Frame: Data will be made available from 1 year after the trial findings are published. This is available for up to 5 years after study completion.
Access Criteria: We will make provision for and consider data sharing requests from bona fide researchers who must abide by the following principles: data will be collected with an high level of quality assurance, data will be held securely with appropriate documentation, data will not be put into the public domain or otherwise shared without explicit ethical review or legal obligation, and they will aim to use any data generated to the maximum public good. These datasets are governed by data usage policies specified by the data controller (UCL). If a conflict exists that severely restricts the analyses that can be undertaken, we would endeavour to support outside researchers by hosting them as visiting workers in our team so that they can access the data. We are committed to complying with the Wellcome Trust Data Sharing Policy. Applications are subject to review by Prof Lovat and Rawen Kader and should be emailed to l.lovat@ucl.ac.uk

RESULTS

PARTICIPANT FLOW:
Groups:
- CADDIE: The endoscopist will be assisted with CADDIE system to detect polyps. The endoscopist will perform optical diagnosis of polyps with the assistance of the CADDIE's polyp characterisation function.
  CADDIE- Computer Aided (AI) Device used in Endoscopy:
  1. CADDIE assisted polyp detection
  2. CADDIE assisted polyp characterisation
Period: Overall Study
Arm/Group | CADDIE | Standard Procedure
Started | 368 | 371
Completed | 306 | 309
Not Completed | 62 | 62

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CADDIE | Standard Procedure | Total
Number analyzed (Participants) | 306 | 309 | 615
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 176 | 201 | 377
  >=65 years | 130 | 108 | 238
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.4 (14.7) | 58.0 (14.8) | 58.7 (14.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 159 | 156 | 315
  Male | 147 | 153 | 300
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity/Race: White British/Irish | 226 | 247 | 473
  Ethnicity/Race: White European | 21 | 16 | 37
  Ethnicity/Race: Mixed race | 3 | 2 | 5
  Ethnicity/Race: South East Asian | 24 | 11 | 35
  Ethnicity/Race: Asian Chinese | 3 | 2 | 5
  Ethnicity/Race: Asian Other | 6 | 3 | 9
  Ethnicity/Race: Black | 4 | 11 | 15
  Ethnicity/Race: Jewish | 1 | 1 | 2
  Ethnicity/Race: Arab | 5 | 6 | 11
  Ethnicity/Race: Other | 13 | 10 | 23
Region of Enrollment [Number; unit: participants]
  United Kingdom | 306 | 309 | 615

OUTCOME MEASURES:

1. Primary Outcome: To Evaluate Whether Using the CADDIE System Improves Endoscopist Detection of Adenomas During Colonoscopy.
Description: The difference in endoscopist ADR between the intervention (CADDIE system) and non-intervention arm.
Time Frame: 30 days
Measure: Number; unit: ADR (% of participants)
Arm/Group | CADDIE | Standard Procedure
Number analyzed (Participants) | 306 | 309
ADR (% of participants) | 33.30 | 25.20

2. Secondary Outcome: Evaluate the Difference in Number of Adenomas Detected Per Colonoscopy Between Intervention and Non-intervention Arm
Description: Compare the difference in the number of adenomas detected per colonoscopy between the intervention and non-intervention arm
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: Adenomas per colonoscopy
Arm/Group | CADDIE | Standard Procedure
Number analyzed (Participants) | 306 | 309
Adenomas per colonoscopy | 0.66 (1.44) | 0.42 (0.98)

3. Secondary Outcome: To Determine Whether the CADDIE Artificial Intelligence System Improves Endoscopic Detection of All Polyps During Colonoscopy
Description: Polyp Detection Rate (including proximal polyp detection rate) in the interventional group compared to the control group.
  - Mean number of polyps detected per colonoscopy in the interventional group compared to the control group.
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: PPC
Arm/Group | CADDIE | Standard Procedure
Number analyzed (Participants) | 306 | 309
PPC | 0.87 (1.59) | 0.63 (1.24)

4. Secondary Outcome: Compare the Accuracy of Endoscopist Optical Diagnosis of Diminutive Polyps When Using the CADDIE System (Intervention Arm) Compared to Without the CADDIE System (Control Arm)
Description: Compare the accuracy of CADDIE against human endoscopist (high confidence diagnoses) for the optical diagnosis of diminutive polyps. Accuracy is defined as true positive and true negative divided by diagnoses total polyps that were optically diagnosed with high confidence.
Time Frame: 30 days
Measure: Number (95% Confidence Interval); unit: % of adenomas correctly diagnosed
Arm/Group | CADDIE | Standard Procedure
Number analyzed (Participants) | 306 | 309
% of adenomas correctly diagnosed | 87.5 [77.6 to 94.1] | 76.7 [64.3 to 86.2]

5. Secondary Outcome: Compare the Accuracy of Endoscopist Optical Diagnosis to Assign Colonoscopy Surveillance Intervals When Using the CADDIE System (Intervention Arm) Compared to Without the CADDIE System (Control Arm)
Description: Compare the accuracy of using CADDIE's optical diagnosis to assign surveillance colonoscopy intervals against using human endoscopist optical diagnosis (high confidence diagnoses) for assigning surveillance colonoscopy intervals.
Time Frame: 30 days
Measure: Number; unit: % pts with correct surveillance interval
Arm/Group | CADDIE | Standard Procedure
Number analyzed (Participants) | 306 | 309
% pts with correct surveillance interval | 90.9 | 87.2

6. Secondary Outcome: Compare the Accuracy of Endoscopist Optical Diagnosis of Diminutive Rectal Polyps When Using the CADDIE System (Intervention Arm) Compared to Without the CADDIE System (Control Arm)
Description: Compare the accuracy of CADDIE against human endoscopist (high confidence diagnoses) for the optical diagnosis of diminutive rectal polyps.
Time Frame: 30 days
Measure: Number (95% Confidence Interval); unit: % of adenomas correctly diagnosed
Arm/Group | CADDIE | Standard Procedure
Number analyzed (Participants) | 306 | 309
% of adenomas correctly diagnosed | 73.3 [44.9 to 92.2] | 53.3 [26.6 to 78.7]

7. Secondary Outcome: Evaluate the Safety of the CADDIE by Recording Occurrence and Severity of Adverse Events.
Description: Safety of the device will be assessed through monitoring of adverse events for 30 days' post-procedure. Adverse events are defined as:
  * Abdominal pain/discomfort.
  * Abdominal bloating.
  * Sedation related aspiration.
  * Bleeding risk.
  * Perforation.
  * Post polypectomy electrocoagulation syndrome.
  * Infection.
Time Frame: 30 days
Measure: Number; unit: AE/SAE
Arm/Group | CADDIE | Standard Procedure
Number analyzed (Participants) | 368 | 371
AE/SAE | 15 | 14

8. Secondary Outcome: Assess Patient Anxiety During the Colonoscopy
Description: Patient response to the question 'How anxious or calm were you during the colonoscopy?' assessed by Likert Scale with 5 options - 1 (Very anxious), 2 (Somewhat anxious), 3 (Neither Anxious nor calm), 4 (Somewhat calm), 5 (Very calm).
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CADDIE | Standard Procedure
Number analyzed (Participants) | 306 | 309
score on a scale | 2.989 (1.193) | 3.061 (1.241)

ADVERSE EVENTS:
Time Frame: Adverse events were recorded for 30 days post-procedure
Arm/Group | CADDIE | Standard Procedure
All-Cause Mortality (participants affected / at risk) | 2/368 | 0/371
Serious Adverse Events (participants affected / at risk) | 5/368 | 1/371
Other Adverse Events (participants affected / at risk) | 10/368 | 13/371
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CADDIE (N=368) | Standard Procedure (N=371)
Re-admission due to fall, mechnical injury (Musculoskeletal and connective tissue disorders) | 1 | 1
Operation unrelated to study design/study device (Surgical and medical procedures) | 1 | 0
Gastrointestinal disorder unrelated to study device (Gastrointestinal disorders) | 1 | 0
Death due to underlying cardiovascular disease (Cardiac disorders) | 1 | 0
Death due to index diagnosis of malignancy unrelated to study design/ study device (General disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CADDIE (N=368) | Standard Procedure (N=371)
Gastrointestinal disorder unrelated to study device (Gastrointestinal disorders) | 2 | 7
Mechanical Injury unrelated to study design/ study device (Musculoskeletal and connective tissue disorders) | 1 | 2
New diagnosis Prostate cancer (Renal and urinary disorders) | 1 | 0
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Headache (Nervous system disorders) | 1 | 0
Electrolyte abnormality (Investigations) | 1 | 0
Irregular heart beat (Cardiac disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Facial pain (Nervous system disorders) | 0 | 1
Pyelonephritis (Renal and urinary disorders) | 1 | 0
AKI (Renal and urinary disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-05): https://cdn.clinicaltrials.gov/large-docs/15/NCT04325815/Prot_SAP_000.pdf